CLINICAL TRIAL: NCT07317921
Title: Validating the Indicator Amino Acid Oxidation Technique for Muscle Outcomes
Brief Title: Validating IAAO for Muscle Outcomes
Acronym: VIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Principal Investigator, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VIM
Record Dates: First submitted 2025-12-18; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Protein Metabolism
Keywords: Muscle biopsy; Protein Metabolism; Stable isotopes; Protein oxidation; Indicator amino acid oxidation; Protein synthesis
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Intervention Model Description: Single group:
  Eight healthy young (18-35 years, 4 females and 4 males) will be subjected to 2 skeletal muscle biopsies, collection of blood and urine samples, and a non-invasive 13CO2 breath-test over a 6.5-hour period while ingesting half-hourly protein beverages with stable isotope tracers. The breath-test is based on the indicator amino acid oxidation (IAAO) method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protein + Stable Isotope Tracer Beverage (Experimental): Participants will consume 12 half-hourly (6 hours) isoenergetic, isonitrogenous beverages containing 0.9g/kg fat-free mass/day protein. Drinks will be enriched with stable isotopes [2H5]Phenylalanine and [1-13C]Phenylalanine, which will respectively allow for determination of muscle protein synthesis and whole-body protein synthesis over the subsequent 6 hours of feeding.
  Interventions: Dietary Supplement: Protein + Stable Isotope Tracer Beverage

INTERVENTIONS:
Dietary Supplement: Protein + Stable Isotope Tracer Beverage — Participants will consume 12 half-hourly (6 hours) isoenergetic, isonitrogenous beverages containing 0.9g/kg fat-free mass/day protein. Drinks will be enriched with stable isotopes [2H5]Phenylalanine and [1-13C]Phenylalanine, which will respectively allow for determination of muscle protein synthesis and whole-body protein synthesis over the subsequent 6 hours of feeding

SUMMARY:
Consuming dietary protein stimulates whole-body and muscle protein synthesis, the latter of which is typically measured using invasive primed constant infusions of stable isotopes with concurrent muscle biopsies. Alternative non-invasive methodologies have been developed (namely the indicator amino acid oxidation (IAAO) technique) to estimate the impact of protein ingestion on whole-body protein synthesis as a proxy for determining dietary protein requirements. Given that the IAAO technique is based on principles of protein metabolism which occur in the liver, it is unclear how representative the IAAO outcomes of whole-body protein synthesis is to skeletal muscle protein synthesis. Validation of the IAAO technique against gold-standard, biopsy-derived measures of muscle metabolism (i.e., muscle protein synthesis) would assist in mitigating the invasiveness of muscle physiology and nutrition research.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be aged 18-35 years old
* Participants will have a BMI within the normal range (i.e., 18.5-24.9) and waist-to-hip circumference ratio of <0.95 for males and <0.8 for circumference for females to ensure homogeneity of the sample population
* Participants are willing to abide by the compliance rules of this study (e.g., abstain from extraneous physical activity 48h prior to session 4
* Self-reported regular menstrual cycle (25-35d) within the last 3 months (female participants)
* Physical activity score of ≥24 units as measured by the Godin leisure time exercise questionnaire

Exclusion Criteria:

* Inability to adhere to any of the compliance rules judged by principal investigator
* Self-reported regular tobacco or illicit drug use (e.g., growth hormone or testosterone)
* Current use of hormonal contraceptives
* Individuals with a history of allergy to local anesthetics (e.g., lidocaine)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Phenylalanine excretion (umol/kg/h) | 6.5 hours
  Rate of whole-body phenylalanine excretion following orally ingested amino acid tracer [1-13C]Phenylalanine determined from the product of breath 13CO2 enrichment and carbon dioxide production rate (VCO2).
Phenylalanine oxidation (umol/kg/h) | 6.5 hours
  Rate of whole-body phenylalanine oxidation following orally ingested amino acid tracer [1-13C]Phenylalanine determined from the correction of phenylalanine excretion by the phenylalanine precursor enrichment via urine enrichment.
Myofibrillar protein synthesis (%/hr) | 6.5 hours
  Rate of myofibrillar fractional synthesis is determined by rate of incorporation of orally ingested tracer [2H5]Phenylalanine into myofibrillar proteins (isolated from skeletal muscle biopsies) and the enrichment of [2H5]Phenylalanine in plasma collected over the 6 hours protein consumption period. Enrichment will be quantified via tandem LC-MS/MS to derive a rate of incorporation over the 6-hour period.
Sarcoplasmic protein synthesis (%/hr) | 6.5 hours
  Rate of sarcoplasmic fractional synthesis is determined by rate incorporation of orally ingested tracer [2H5]Phenylalanine into sarcoplasmic (ie., soluble) proteins (isolated from skeletal muscle biopsies) and the enrichment of [2H5]Phenylalanine in plasma collected over the 6 hours protein consumption period. Enrichment will be quantified via tandem LC-MS/MS to derive a rate of incorporation over the 6-hour period.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Moore, Ph.D, Principal Investigator — University of Toronto, Faculty of KPE
Locations (1):
- Kinesiology & Physical Education, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided